CLINICAL TRIAL: NCT02655952
Title: Phase Ib Dose Escalating Study to Evaluate the Safety, Tolerability and Pharmacodynamic Response of Foxy-5 in Patients With Metastatic Breast-, Colon- or Prostate Cancer
Brief Title: Dose Escalating Study of Foxy-5 in Breast-, Colon- or Prostate Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: WntResearch AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMR-3164
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Breast Cancer; Metastatic Colon Cancer; Metastatic Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Prostatic Neoplasms | interventions — Foxy-5 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Foxy-5 (Experimental): Slow infusion of lyophilised and reconstituted Foxy-5 three times weekly for three weeks.
  There will be a maximum of 8 dose cohorts. Cohorts 1-4 will be conducted in the United Kingdom and Denmark whereas cohorts 5-8 will only be conducted in Denmark. As doses in cohort 1 and 2 have been investigated in the previous phase I study, cohorts 1+2 and 3 can be run in parallel with dose escalation approved by the DSMB at all times.
  DK+UK: Cohort 1: 0.8 mg/kg DK+UK: Cohort 2: 1.3 mg/kg DK+UK: Cohort 3: 1.8 mg/kg DK+UK: Cohort 4: 2.3 mg/kg DK only: Cohort 5: 3.0 mg/kg DK only: Cohort 6: 4.0 mg/kg DK only: Cohort 7: 5.3 mg/kg DK only: Cohort 8: 7.0 mg/kg
  Interventions: Drug: Foxy-5

INTERVENTIONS:
Drug: Foxy-5

SUMMARY:
The Wnt proteins belong to a family of proteins that have been demonstrated to play a role in the formation and dissemination of tumours. The present project focuses on the critical role of the Wnt-5a protein in the pathobiological processes that lead to metastatic cancer disease.

WntResearch has identified a formylated 6 amino acid peptide fragment, named Foxy-5, which mimick the effects of Wnt-5a to impair migration of epithelial cancer cells and thereby acting anti-metastatic.

The aim of the first clinical phase I study was to establish the recommended dose for a clinical phase II study and enable further development of Foxy-5 as a first in class anti-metastatic cancer drug. The study did not see any DLTs and therefore failed to reach maximum tolerated dose (MTD); no recommended phase II dose (RP2D) could therefore be established based on toxicity. The aim of this study is to continue to establish the safety profile of Foxy-5 in higher doses, and determine the RP2D for later stage development based on any observed DLT's/MTD and further analysis of the pharmacodynamic profile of Foxy-5 to determine the biological response dose (BRD).

ELIGIBILITY:
Inclusion Criteria:

* Males and females of at least 18 years of age

  * Histologically/cytologically documented diagnosis of metastatic breast, colon or prostate cancer, refractory to standard therapy or for which no curative therapy exists
  * Must have an evaluable tumour appropriate for biopsy as determined by the Investigator.
  * Loss of or reduced Wnt-5a protein expression in primary or metastatic tumour cells, characterised by IHC analysis
  * Eastern Cooperative Oncology Group (ECOG) performance status of <= 1
  * Life expectancy of at least 3 months
  * Unresectable disease, i.e. the metastases cannot be surgically removed with a curative intent

    * 4 weeks must have elapsed since the patient has received any other IMP
    * 4 weeks must have elapsed since the patient has received any anti cancer treatment; including radiotherapy (except for single dose of palliative radiotherapy), cytotoxic chemotherapy, biologic agents or targeted therapy
    * 2 weeks must have elapsed since any prior surgery or therapy with bone marrow stimulating factors
  * Adequate haematological functions as defined by:
  * Absolute neutrophil count >= 1.5 10E9/L
  * Platelets >= 100 10E9/L
  * Hemoglobin >= 5.6 mmol/L
  * Adequate hepatic function as defined by:
  * Total bilirubin <= 1.5 x the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) <= 2.5 x ULN*
  * Alanine aminotransferase (ALT) <= 2.5 x ULN*

    * For patients with liver metastasis adequate hepatic function is defined by AST <= 5 x ULN and ALT <= 5 ULN.
  * Adequate renal function as defined by Serum creatinine <= 1,5 x ULN
  * Patients in active anti-coagulating treatment must be evaluated according to local standards on the discretion of the Investigator..
  * Provision of written informed consent
  * Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
  * Sexually active males and females of child-producing potential, must use adequate contraception (intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release) or diaphragm always with spermicidal jelly and a male condom) for the study duration and at least six months afterwards

Exclusion Criteria:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease)

  * Any active infection requiring antibiotic treatment
  * Known infection with human immunodeficiency virus (HIV) or hepatitis virus
  * Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or symptomatic arrhythmias currently requiring medication
  * Known or suspected active central nervous system (CNS) metastasis. (Patients stable 8 weeks after completion of treatment for CNS metastasis are eligible)
  * Impending or symptomatic spinal cord compression or carcinomatous meningitis
  * Requiring immediate palliative surgery and/or radiotherapy(except for a single dose of palliative radiotherapy)
  * Pre-existing neuropathy, i.e., Grade >2 neuromotor or neurosensory toxicity
  * Participation in other clinical studies within 4 weeks of first dose of study treatment
  * Previous exposure to Foxy-5
  * History of severe allergic or hypersensitive reactions to excipients
  * Pregnant or breastfeeding women
  * Active and/or within the last 5 years histologically confirmed diagnosis of malignant melanoma, gastric cancer, pancreatic cancer, lung cancer or nasopharyngeal cancer
  * Severe or uncontrolled chronic or uncontrolled systemic disease (e. g. severe respiratory or cardiovascular disease)
  * Other medications or conditions that in the Investigator's opinion would contraindicate study participation of safety reasons or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Presence of Dose Limiting Toxicities (DLTs). | 6 month
  The number of adverse events along with the results of vital sign measurements, physical examinations, and clinical laboratory tests will be used to determine the safety and tolerability profile of Foxy-5

SECONDARY OUTCOMES:
Genome wide mRNA gene expression in tumour biopsies and blood (buffy coat) | Tumour biopsies obtained prior to day 1 and on day 12 and 19
  Determination of the biological response dose (BRD) based on the alterations in the exploratory biomarkers during treatment with Foxy-5
Wnt-5a protein expression and hematoxylin-eosin (HE) staining of tumour biopsies | Tumour biopsies obtained prior to day 1 and on day 12 and 19
  Determination of the biological response dose (BRD) based on the alterations in the exploratory biomarkers during treatment with Foxy-5
Numbers of circulating tumour cells (CTCs) in blood | Blood sample obtained prior to day 1 and on day 12 and 19
  Determination of the biological response dose (BRD) based on the alterations in the exploratory biomarkers during treatment with Foxy-5
Maximum tolerated dose (MTD) | 6 month
  Determined as the dose preceding the dose at which two or more patients have experienced DLTs. Assessment of adverse events and laboratory abnormalities
Area under the plasma concentration curve (AUC) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Bioavailability (F) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Half life (T½) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Absorption rate Constant (tmax) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Volume of distribution (V) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Clearance (C) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Extraction Ratio (E) of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)
Hepatic and Renal Clearance of Foxy-5 | immediately prior to treatment, at 0, 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion.
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Tine Mølvadgaard, M.Sc.Pharm, Study Director — Smerud Medical Research Denmark
Locations (4):
- Denmark (3):
  - Clinical Research Department, Oncology, Rigshospitalet, Copenhagen
  - Onkologisk Afdeling R, Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- NCCC, Freeman Hospital, Newcastle, Newcastle Upon Tyne, United Kingdom